CLINICAL TRIAL: NCT05410977
Title: Detection of Colorectal Cancer or Advanced Neoplasia by Stool DNA in Lynch Syndrome: CORAL Study
Brief Title: Collecting Blood and Stool Samples to Detect Colorectal Cancer or Advanced Neoplasia in Lynch Syndrome Patients
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CORAL; NCI-2022-02032 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-010010 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Carcinoma; Lynch Syndrome
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, record review): Patients undergo collection of blood and stool samples no more than 90 days prior to or between 7-90 days after standard of care colonoscopy or flexible sigmoidoscopy. Patients' medical records are also reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and stool samples
Other: Electronic Health Record Review — Medical records reviewed

SUMMARY:
This study collects blood and stool samples from patients with suspected or diagnosed Lynch syndrome to evaluate a deoxyribonucleic acid (DNA) screening technique for the detection of colorectal cancer in Lynch syndrome patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the sensitivity and specificity of the multitarget stool DNA (mt-sDNA) 2.0 test, for colorectal neoplasia in patients with Lynch syndrome.

SECONDARY OBJECTIVE:

I. Develop a biorepository of samples (stool and blood) from patients with Lynch syndrome and early onset (< 50 years old) colorectal cancer.

OUTLINE:

Patients undergo collection of blood and stool samples no more than 90 days prior to or between 7-90 days after standard of care colonoscopy or flexible sigmoidoscopy. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* Individuals diagnosed with Lynch syndrome (mutation in MLH1, MSH2, MSH6, PMS2, EPCAM) or suspected Lynch syndrome or individuals diagnosed with early onset colorectal cancer (CRC) (< 50 years old)
* Colonoscopy/flexible sigmoidoscopy (flex sig) scheduled +/- 90 days from sample collection
* Patient has agreed to participate and has signed the study consent form

Exclusion Criteria:

* Patient has known cancer (stage I-IV) 5 years prior to current sample collection (not including basal cell or squamous cell skin cancers; if patient has not been seen or if information is not available, the patient is eligible)
* Patient has received chemotherapy class drugs for the treatment of cancer in the 5 years prior to current sample collection
* Patient has had any abdominal radiation therapy prior to current sample collection
* Patient had therapy to the target lesion with intent to completely remove or debulk the lesion prior to sample collection [examples include snare polypectomy, endoscopic mucosal resection (EMR), endoscopic submucosal dissection (ESD), surgical resection, trans anal excision]
* Patient has prior diagnosis of non-lynch hereditary colon cancer syndrome [familial adenomatous polyposis (FAP), MUTYH-associated polyposis (MAP), Peutz-Jeghers syndrome (PJS), juvenile polyposis syndrome (JPS), PTEN, POL]
* ADDITIONAL STOOL EXCLUSIONS:
* Bowel prep < 7 days prior to stool collection
* Oral or rectal contrast given within 7 days prior to stool collection
* Removal of more than 50% of colon or presence of ileostomy
* Enteral feeds or total parenteral nutrition (TPN)
* Diagnosis of inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with Lynch syndrome or suspected Lynch syndrome or early onset colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of multitarget stool deoxyribonucleic acid (mt-sDNA) 2.0 test to detect colorectal neoplasia | Up to 4 years
  Results of the mt-sDNA 2.0 test will be correlated with pathology findings of patients undergoing colonoscopy to determine sensitivity of the mt-sDNA 2.0 test
Specificity of mt-sDNA 2.0 test to detect colorectal dysplasia | Up to 4 years
  Results of the mt-sDNA 2.0 test will be correlated with pathology findings of patients undergoing colonoscopy to determine specificity of the mt-sDNA 2.0 test

CONTACTS AND LOCATIONS:
Overall Officials: Niloy Jewel Samadder, M.D., Principal Investigator — Mayo Clinic
Locations (9):
- United States (9):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of California San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Center, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials